CLINICAL TRIAL: NCT02183155
Title: A Double Blind, Randomized, Parallel Group Trial to Compare the Effect of Three Doses of Meloxicam Tablets (7.5, 15 and 30 mg) With Placebo on Bleeding Time in Healthy Subjects; With Extended-release Indomethacin Capsules 75 mg (Open-label) as an Active Control to Assess Trial Sensitivity.
Brief Title: Effect of Meloxicam Tablets on Bleeding Time in Healthy Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107.236
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (5):
- Meloxicam - low (Experimental)
  Interventions: Drug: Meloxicam - low
- Meloxicam - medium (Experimental)
  Interventions: Drug: Meloxicam - medium
- Meloxicam - high (Experimental)
  Interventions: Drug: Meloxicam - high
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Extended-release indomethacin (Active Comparator)
  Interventions: Drug: Extended-release indomethacin

INTERVENTIONS:
Drug: Meloxicam - low
  Arms: Meloxicam - low
Drug: Meloxicam - medium
  Arms: Meloxicam - medium
Drug: Meloxicam - high
  Arms: Meloxicam - high
Drug: Placebo
  Arms: Placebo
Drug: Extended-release indomethacin
  Arms: Extended-release indomethacin

SUMMARY:
The primary purpose of this study was to evaluate the effect of meloxicam tablets (7.5, 15 mg and 30 mg) with meloxicam placebo. Extended-release indomethacin capsules (75 mg) was an active control to assess trial sensitivity on bleeding time in healthy subjects. The secondary aim of this study was to assess effects of treatment on other platelet function and coagulation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between the ages of 18 and 55 years
* Negative urine pregnancy test on Day1 for females of childbearing potential
* Weight within +/- 20 percent of ideal weight according to the Metropolitan Life Height and Weight chart
* Willing and able to cooperate with the investigator and his/her staff
* Written informed consent in accordance with GCP (Good Clinical Practice) and local legislation

Exclusion Criteria:

* Any finding, medical condition or dietary restriction that, in the investigator's opinion, may interfere with optimal participation in the study or produce a significant risk to the subject
* In the opinion of the investigator, the subject has any disease or condition that may result in altered absorption, excess accumulation, or impaired metabolism or excretion of the trial medications
* A known or suspected hypersensitivity to any of the trial medications or their excipients or any other NSAIDs (Non-Steroid Anti-Inflammatory Drug)
* A history of gastrointestinal ulcer, perforation or bleeding
* A history of cerebrovascular bleeding or any other bleeding disorder
* Women of childbearing potential not using adequate contraception (e.g, intrauterine device, contraceptive pills, Depo-Provera® implant, barrier device) for at least 3 months prior to, and for the duration of trial participation. It should be noted that NSAIDs may interfere with the effectiveness of intrauterine devices
* History of bronchial asthma
* Use of any medications that might influence the results of the trial
* Use of anticoagulants, including warfarin, heparin, ticlopidine, clopidogrel or aspirin
* Any laboratory value outside the normal range that is considered clinically significant by the investigator. In addition, subjects with the following specific laboratory values will not be allowed:

  * A serum creatinine concentration at baseline > 1.5 mg/dl
  * SGOT (serum glutamic-oxaloacetic transaminase) or SGPT (serum glutamic-pyruvic transaminase) liver enzymes results at baseline > 1.5 times the upper limit of normal
  * A hemoglobin concentration < 10.5 g/dl
  * A white cell count < 3500/mm³
  * A platelet < 100,000/mm³ or a documented abnormal bleeding time, platelet aggregation, thromboxane B2 synthesis, thromboplastin time (PT) or activated partial thromboplastin time (APTT)
* Inability to refrain from smoking on testing days
* Participation in another trial with an investigational drug within 30 days of entering the trial
* Subjects with increased keloid formation
* Previous surgery of the gastrointestinal tract (except appendectomy)
* Participation in excessive physical activities (≤ 5 days prior to administration)
* Current drug or alcohol abuse
* Small or difficult to locate arm veins that would impair the clinician's ability to draw blood samples
* Homeopathic medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2000-05; Primary Completion 2000-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in bleeding time | up to 6 hours post-dose at day 8

SECONDARY OUTCOMES:
Change from baseline in platelet aggregation | up to 6 hours post-dose at day 8
Change from baseline in Platelet thromboxane B2 synthesis (TXB2 synthesis) | up to 6 hours post-dose at day 8
Change in Thromboplastin Time (PT) | up to 6 hours post-dose at day 8
Change in Activated Partial Thromboplastin Time (APTT) | up to 6 hours post-dose at day 8
Change in Platelet Count | up to 6 hours post-dose at day 8
Change in Leucocyte Activation | Day 1 and 6 hours post-dose at day 8
Plasma levels of meloxicam | pre-dose, 3 and 6 hours post-dose at day 8
Plasma levels of indomethacin | pre-dose, 3 and 6 hours post-dose at day 8
Number of patients with adverse events | up to 8 days